CLINICAL TRIAL: NCT02935790
Title: A Phase 1b Study of the Selective HDAC6 Inhibitor ACY-241 in Combination With Ipilimumab and Nivolumab in Patients With Unresectable Stage III or Stage IV Melanoma
Brief Title: Selective HDAC6 Inhibitor ACY-241 in Combination With Ipilimumab and Nivolumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Syneos Health (Other); ApoCell, Inc. (Industry); Celerion (Industry); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-ST-204
Record Dates: First submitted 2016-05-03; First posted 2016-10-18 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Malignant Melanoma
Keywords: unresectable; melanoma
MeSH Terms: conditions — Melanoma | interventions — citarinostat; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACY-241 combo with Ipi and Nivo (Experimental): ACY-241 in Combination with Ipilimumab and Nivolumab
  Interventions: Drug: ACY-241; Drug: nivolumab; Drug: ipilimumab

INTERVENTIONS:
Drug: ACY-241 — tablet
  Other Names: HDAC6 Inhibitor
Drug: nivolumab — infusion
  Other Names: OPDIVO
Drug: ipilimumab — infusion
  Other Names: YERVOY

SUMMARY:
Determine the safety, tolerability, dose-limiting toxicities (DLTs), maximum tolerated dose (MTD), and recommended Phase 2 dose (RP2D) of ACY-241 in combination with ipilimumab and nivolumab in patients with unresectable Stage III/Stage IV melanoma.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, dose-escalation cohort study. The study will consist of a dose escalation assessment of the safety and tolerability of ACY-241 administered concurrently in combination with ipilimumab and nivolumab to patients with advanced melanoma. Treatment will be divided into induction and maintenance phases.

Determine the safety, tolerability, dose-limiting toxicities (DLTs), maximum tolerated dose (MTD), and recommended Phase 2 dose (RP2D) of ACY-241 in combination with ipilimumab at 1 mg/kg and nivolumab at 3 mg/kg every 3 weeks for 4 doses each during a 12-week induction period, then administered with nivolumab at a flat dose of 240 mg every 2 weeks in maintenance for up to 1 year in patients with unresectable Stage III/Stage IV melanoma.

It is anticipated that this clinical study will enable selection of the RP2D and dose schedule of this 3-drug combination for further clinical testing. The trial will include an assessment of the pharmacodynamic activity of ACY-241.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed and dated an Institutional Review Board/Independent Ethics Committee -approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal patient care
2. Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study.
3. All patients must be either Stage IIIb/c or Stage IV according to the American Joint Committee on Cancer (AJCC) (7th edition) and have histologically-confirmed melanoma that is felt to be surgically unresectable in order to be eligible. Please refer to the AJCC Cancer Staging Manual, 7th edition for a description of tumor, lymph node, metastasis and staging.

   * All melanomas, except ocular/uveal melanoma, regardless of primary site of disease will be allowed; mucosal melanomas are eligible.
   * Patients must not have received prior anticancer treatment for metastatic disease (for example, but not limited to, systemic, local, radiation, radiopharmaceutical).

     -Exceptions: Surgery for melanoma and/or postresection brain radiotherapy (RT) if central nervous system (CNS) metastases and/or prior treatment with adjuvant interferon (IFN) (as described in Exclusion Criterion 2).
   * All patients must have their disease status documented by a complete physical examination and imaging studies within 4 weeks prior to the first dose of study drug. Imaging studies must include computerized tomography (CT) scan of neck, chest, abdomen, pelvis, and all known sites of resected disease in the setting of Stage IIIb/c or Stage IV disease, and brain magnetic resonance imaging ([MRI], brain CT allowable if MRI is contraindicated).
   * The complete set of baseline radiographic images must be available before treatment initiation.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
5. Tumor tissue from the resected site of disease must be provided for biomarker analyses
6. Prior treated CNS metastases must be without MRI evidence of recurrence for at least 4 weeks after treatment. Patients must be off immunosuppressive doses of systemic steroids (≥ 10 mg/day prednisone or equivalent) for at least 14 days prior to study drug administration, and must have returned to neurologic baseline status postoperatively.

   • The 4-week period of stability is measured after the completion of the neurologic interventions (ie, surgery and/or radiation).
7. In addition to neurosurgery to treat CNS metastases, adjuvant radiation after the resection of CNS metastasis is allowed. Immunosuppressive doses of systemic steroids (doses ≥ 10 mg/day prednisone or equivalent) must be discontinued at least 14 days before study drug administration.
8. Prior surgery that required general anesthesia must be completed at least 4 weeks before study drug administration. Surgery requiring local/epidural anesthesia must be completed at least 72 hours before study drug administration.
9. All baseline laboratory requirements will be assessed and should be obtained within 14 days of first dose of study drug. Screening laboratory values must meet the following criteria:

   * White blood cells ≥ 2000/µL
   * Neutrophils ≥ 1500/µL
   * Platelets ≥ 100 × 10³/µL
   * Hemoglobin ≥ 9.0 g/dL
   * Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance > 40 mL/minute (using Cockcroft/Gault formula)
10. Patient Re-enrollment: This study permits the re-enrollment of a patient that has discontinued the study as a screen failure (ie, patient has not been dosed/has not been treated). If re-enrolled, the patient must be re-consented.
11. Males and females ≥ 18 years of age.
12. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin hormone) within 24 hours prior to the start of study drug.
13. Women must not be breastfeeding.
14. Women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of study drug plus 30 days (duration of ovulatory cycle). The half-lives of nivolumab and ipilimumab is up to 25 days and 18 days, respectively. Given the blinded nature of this study, WOCBP should therefore use an adequate method to avoid pregnancy for a total of 23 weeks posttreatment completion.
15. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half lives of the study drug(s) plus 90 days (duration of sperm turnover). The half-lives of nivolumab and ipilimumab are up to 25 days and 18 days, respectively. Given the blinded nature of this study, men should therefore use an adequate method of contraception for a total of 31 weeks posttreatment completion.
16. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing as described in this section.

Investigators shall counsel WOCBP and male patients who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and male patients who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

Exclusion Criteria:

1. Patients with carcinomatosis meningitis or a history of ocular/uveal melanoma are excluded.
2. Patients with previous nonmelanoma malignancies are excluded unless a complete resection or remission was achieved at least 2 years prior to study entry and no additional therapy is required or anticipated to be required during the study period (exceptions include, but are not limited to, nonmelanoma skin cancers, in situ bladder cancer, in situ gastric cancer or gastrointestinal stromal tumor, in situ colon cancers, in situ cervical cancers/dysplasia, or breast carcinoma in situ).
3. Patients with active, known, or suspected autoimmune disease. Patients with type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll. For any cases of uncertainty, it is recommended that the Principal Investigator be consulted prior to signing informed consent.
4. Patients with a condition requiring systemic treatment with either corticosteroids (≥ 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
5. Prior therapy for melanoma with the following exceptions which are allowed: 1) surgery for the melanoma lesion(s), 2) adjuvant RT after neurosurgical resection for CNS lesions, and 3) prior adjuvant IFN (see qualifier below). Specifically, patients who received prior therapy with anti-PD-1, anti PD L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T cell costimulation or checkpoint pathways) are not eligible.

   • Prior treatment with adjuvant IFN is allowed if completed ≥ 3 months prior to treatment.
6. Treatment directed against the melanoma (eg, chemotherapy, targeted agents, biotherapy, limb perfusion) that is administered after a prior complete resection other than adjuvant radiation after neurosurgical resection and IFN for resected melanoma.
7. Previous therapy with histone deacetylase inhibitor.
8. Any of the following laboratory abnormalities:

   * ANC < 1,500/µL
   * Platelet count < 100,000/µL
   * Hematologic growth factors are not allowed at screening or during the first cycle of treatment
   * Hemoglobin < 9 g/dL (< 5.5 mmol/L; previous red blood cell transfusion is permitted)
   * Creatinine > 1.5 × ULN
   * AST or ALT > 2.5 × ULN. For patients with liver metastasis, AST or ALT > 5 × ULN
   * Serum total bilirubin > 1.5 mg/dL or > 3 × ULN for patients with hereditary benign hyperbilirubinemia
9. Corrected QT interval (QTc) using Fridericia's formula value > 480 msec at screening; family or personal history of long QTc syndrome or ventricular arrhythmias including ventricular bigeminy at screening; previous history of drug induced QTc prolongation or the need for treatment with medications known or suspected of producing prolonged QTc intervals on electrocardiogram (ECG).
10. Congestive heart failure (New York Heart Association Class III or IV), myocardial infarction within 12 months before starting study treatment, or unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris.
11. Any serious or uncontrolled medical disorder or active infection that, in the opinion of the Investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the patient to receive protocol therapy.
12. Any positive test result for hepatitis B virus or hepatitis C virus indicating acute or chronic infection.
13. Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome.
14. History of Grade ≥ 3 allergy to human monoclonal antibodies.
15. Prisoners or patients who are involuntarily incarcerated.
16. Patients who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
17. Pregnant or nursing women.
18. Psychological, familial, sociological, or geographical conditions that potentially hamper compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Number of Dose Limiting Toxicities defining the MTD | 12 months

SECONDARY OUTCOMES:
Percentage of Patients with ORR based on RECIST 1.1 change from baseline by CT or MRI measurements | 12 months
Percentage of Patients with ORR based on irRC change from baseline by CT or MRI measurements | 12 months
Maximum observed concentration (Cmax) of ACY-241 administered in combination with ipilimumab and nivolumab | 12 months
trough concentrations of ACY-241 administered in combination with ipilimumab and nivolumab | 12 months

OTHER OUTCOMES:
Exploratory: Pharmacodynamic changes in biomarkers (to be determined) pre-dose versus post-dose in peripheral blood and tumor tissue | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Weber, Principal Investigator — Laura and Isaac Perlmutter Cancer Center, NYU Langone Medical Center; Elizabeth Buchbinder, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided